CLINICAL TRIAL: NCT01024712
Title: Paclitaxel/Carboplatin Combined With Intermittent Gefitinib in Patients With Untreated Advanced Non-small Cell Lung Cancer: A Phase Ⅱa Trial
Brief Title: Paclitaxel, Carboplatin, and Gefitinib in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CIH-CAMS-CHL-020; CDR0000643743 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-12

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Gefitinib; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: gefitinib
Drug: paclitaxel
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving paclitaxel and carboplatin together with gefitinib may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving paclitaxel and carboplatin together with gefitinib and to see how well it works in treating patients with Stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy, in terms of overall response, and safety of paclitaxel and carboplatin in combination with intermittent gefitinib in patients with advanced nonsquamous non-small cell lung cancer.

Secondary

* Determine the disease-control rate in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the progression-free and overall survival of patients treated with this regimen.

OUTLINE: Patients receive paclitaxel IV on day 1, carboplatin IV on day 2, and oral gefitinib once daily on days 8-17. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. After completion of 4 courses, patients with complete response or partial response may continue maintenance therapy comprising oral gefitinib once daily in the absence of disease progression or unacceptable toxicity.

Patients complete the Functional Assessment of Cancer Therapy-Lung (FACT-L) at baseline, during study treatment, and after completion of study treatment for quality-of-life study.

After completion of study treatment, patients are followed every 2 months for 2 years and then every 4 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * No squamous cell carcinoma
* Untreated Stage IIIB or IV disease not suitable for surgery or radiotherapy OR patients with postoperative recurrence who had never been treated by chemotherapy
* No history of smoking or light smoking (< 10 packs a year and smoking abatement ≥ 15 years)
* At least 1 measurable tumor mass (length > 1.5 cm and width > 1.0 cm)
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count ≥ 2 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* ALT and AST ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤1.5 times ULN
* Serum creatinine normal
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignant tumors within the past year except for basal cell or squamous cell carcinoma of the skin, or in situ malignant cancer that has been completely resected
* No history of allergic reaction to any component of the drugs in this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 1 month since prior investigational drugs or medical devices
* No prior chemotherapy or radiotherapy for this tumor
* No concurrent liposomal paclitaxel
* No other concurrent antitumor therapy (e.g., radiotherapy or surgical treatment)
* No other concurrent anticancer chemotherapy drugs or anticancer Chinese herbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
Overall-response rate

SECONDARY OUTCOMES:
Disease-control rate
Safety
Quality of life
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute Hospital, Chinese Academy of Medical Sciences, Beijing, China